CLINICAL TRIAL: NCT01395316
Title: Alemtuzumab on Surrogate Markers of Disease Activity and Repair Using Advanced MRI Measures in Subjects With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-490B
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental): Single arm, single cohort study, all subjects will be dosed with alemtuzumab.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — 10 mg/ml alemtuzumab intravenous infusion, sterile clear, colorless solution. dosage: 2 cycles. Month 0 dosed over 5 consecutive days: month 12 dosed over 3 consecutive days.
  Other Names: CamPath; MabPath

SUMMARY:
The MRI study is designed to identify possible mechanisms by which alemtuzumab acts to protect the brain from inflammation and how it may enhance repair through remyelination.

DETAILED DESCRIPTION:
To identify specific changes in T cell subsets and functions in Relapsing Remitting Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria

1. Signed, informed consent form (ICF)
2. Age 18 to 50 years old (inclusive) as of signing the ICF
3. Diagnosis of MS per update of McDonald criteria, and cranial MRI scan demonstrating white matter lesions attributable to MS within 10 years of screening
4. Onset of MS symptoms (as determined by a neurologist) within 15 years of screening
5. EDSS score 0.0 to 5.0 (inclusive)
6. >=2 MS attacks (first episode or relapse) occurring in the 24 months prior to screening, with >=1 attack in the 12 months prior to screening, with objective neurological signs confirmed by a physician
7. Subjects previously enrolled and randomized to interferon beta 1a in the CARE-MS 323 and 324 studies, and who will be treated with Alemtuzumab through the CARE-MS extension study will be eligible to participate in the immunology and MRI studies of this protocol.

Exclusion Criteria

1. Received prior therapy for MS other than corticosteroids within 28 days of screening; e.g., interferons, IV immunoglobulin, and glatiramer acetate
2. Exposure to natalizumab within 6 months of screening
3. Any prior exposure to mitoxantrone, mycophenolate mofetil, azathioprine, cladribine, cyclophosphamide, cyclosporine A, methotrexate, rituximab, or any other immunosuppressive agent other than systemic corticosteroid treatment
4. Has any progressive form of MS
5. History of malignancy (exception for basal cell skin carcinoma)
6. Previous hypersensitivity reaction to other immunoglobulin product
7. Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
8. CD4+, CD8+, or CD19+ (i.e., absolute CD3+CD4+, CD3+CD8+, or CD19+/mm3) count <LLN at Screening; if abnormal cell count(s) return to within normal limits, eligibility may be reassessed
9. Seropositivity for human immunodeficiency virus (HIV)
10. Significant autoimmune disease (e.g, immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders; vasculitis; inflammatory bowel disease; severe psoriasis)
11. Presence of anti-thyroid stimulating hormone (TSH) receptor (TSHR) antibodies
12. Active infection, e.g, deep-tissue infection, that the Investigator considers sufficiently serious to preclude study participation
13. Latent tuberculosis unless effective anti-tuberculosis therapy has been completed, or active tuberculosis. Patients will be assessed for this risk based on a screening questionnaire.
14. Infection with hepatitis B virus or hepatitis C virus
15. Of childbearing potential with a positive serum pregnancy test
16. Unwilling to agree to use a reliable and acceptable contraceptive method throughout the study period
17. Major psychiatric disorder that is not adequately controlled by treatment
18. Epileptic seizures that are not adequately controlled by treatment
19. Major systemic disease or other illness that would, in the opinion of the Investigator, compromise patient safety or interfere with the interpretation of study results
20. Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study
21. Confirmed platelet count < the lower limit of normal (LLN) of the evaluating laboratory at Screening or documented at <100,000/uL within the past year on a sample without clumping
22. Prior history of invasive fungal infections
23. Cervical high risk human papillomavirus (HPV) positivity or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS). The patient may be eligible after the condition has been effectively treated (eg, follow-up HPV test is negative or cervical abnormality has been treated).
24. Seropositive for Trypanosoma cruzi or the Human T-lymphotropic virus type I or type II (HTLV-I/II) (testing required in endemic regions only)
25. Any other illness or infection (latent or active) that, in the Investigator's opinion, could be exacerbated by alemtuzumab treatment
26. Any hepatic or renal function value grade 2 or higher at Screening, with the exception of hyperbilirubinemia due to Gilbert's syndrome. See Table below, drawn from the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE), published 09 August 2006

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Javed, MD, Principal Investigator — University of Chicago

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 8
Completed | 5
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — poor MRI quality | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Diffusion and Myelin Fraction Water Changes on Magnetic Resonance Imaging (MRI)
Description: Changes in normal appearing white matter from baseline through month 24.
  The MRI is designed to identify possible mechanisms by which alemtuzumab acts to protect the brain from inflammation and how it may enhance repair through remyelination.
Time Frame: Baseline to Month 24
Measure: Mean (Standard Deviation); unit: percent Change
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 5
percent Change | -2.06 (0.01)

ADVERSE EVENTS:
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=8)
Hypothyroidism (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes